CLINICAL TRIAL: NCT05172102
Title: Effect of Breathing Exercise on Chest Expansion, Quality of Life and Lung Function on Post Covid-19 Patient: A Randomized Controlled Trial
Brief Title: Quality of Life and Lung Function on Post Covid-19 Patient
Acronym: Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Maged Basha, Principal Investigator, Assistant Professor of physical therapy, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-04-Q-001
Record Dates: First submitted 2021-12-25; First posted 2021-12-29 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Breathing Exercises; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Will receive diaphragmatic breathing with pursed lips as (breathing exercise), They will instruct to perform 3 different conditions will be registered: (1) 6 min of quiet breathing (3 sets of 2 min each), defined as spontaneous breathing pattern; (2) 6 min of diaphragmatic breathing (3 sets of 2 min each); and (3) 6 min of diaphragmatic breathing plus pursed-lips breathing (3 sets of 2 min each).
  For aerobic exercises: Will include the following exercises: walking, cycling, running and intermittent running. The exercises will perform for 18-60 minutes for 1-2 sets per week.
  For resistance exercises: Will include the following 8 exercises: shoulder press, biceps curl, triceps curl, bench press, leg squats, leg press, leg curl and toe raise. The exercises will perform for 60 minutes for 2-3 sets per week.
  Interventions: Other: breathing exercise, Aerobic exercises
- control group (No Intervention): not receiving any exercises

INTERVENTIONS:
Other: breathing exercise, Aerobic exercises — 6 min of quiet breathing (3 sets of 2 min each), 6 min of diaphragmatic breathing (3 sets of 2 min each), 6 min of diaphragmatic breathing plus pursed-lips breathing (3 sets of 2 min each).
  Other Names: resistance exercises
  Arms: study group

SUMMARY:
Gaining a greater understanding of how the breathing exercise combined with aerobic and strengthening exercises will affects lung function and quality of life in post covid-19 persons

DETAILED DESCRIPTION:
this will improve exercise prescription guidelines relevant to this post covid-19. Therefore, the purpose of this work was determining the effect of breathing exercise combined with aerobic and strengthening exercises in improve chest expansion, lung function and quality of life in post covid-19 persons.

ELIGIBILITY:
Inclusion Criteria:

* Female. Age from 20 to 30 years old. - Body mass index (BMI) 19 to 24 kg/m2.- Non-smoker- Recovered from COVID-19 over the past 12 months. - They are experiencing mild to moderate symptoms without any complications. -
* Able to use online communication programs.

Exclusion Criteria:

* - Anyone who does regular physical exercise.
* history of acute illness, asthma, pulmonary fibrosis, hypertension, diabetes disease.
* hypoxemia in rest.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life, Medical Outcomes Study short-form (SF-36) | at baseline
  assessed using the Short Form-36 (SF-36). The SF-36 scale had 8 dimensions, and each dimension was converted into a percentage score.
Health-related quality of life, Medical Outcomes Study short-form (SF-36) | after 6 weeks
  assessed using the Short Form-36 (SF-36). The SF-36 scale had 8 dimensions, and each dimension was converted into a percentage score.
Respiratory function measurement | at baseline
  assessed by a spirometer. The following parameters related to respiratory function will be measured: (1) forced expiratory volume in 1 second (FEV1); (2) forced vital capacity (FVC).
Respiratory function measurement | after 6 weeks
  assessed by a spirometer. The following parameters related to respiratory function will be measured: (1) forced expiratory volume in 1 second (FEV1); (2) forced vital capacity (FVC).

SECONDARY OUTCOMES:
Chest expansion measurement | at baseline
  measured with a tape measure at 2 different levels of the rib cage. Measurements will be taken at the maximal inspiration and expiration
Chest expansion measurement | after 6 weeks
  measured with a tape measure at 2 different levels of the rib cage. Measurements will be taken at the maximal inspiration and expiration
Exercise endurance measurement | at baseline
  measured by the 6-min walk test (6MWT), is the distance one walks within 6 min
Exercise endurance measurement | after 6 weeks
  measured by the 6-min walk test (6MWT), is the distance one walks within 6 min

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Mahmoud, PhD, Study Director — Qassim University
Locations (1):
- College of medical rehabilitation, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study is available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Result] Liu K, Zhang W, Yang Y, Zhang J, Li Y, Chen Y. Respiratory rehabilitation in elderly patients with COVID-19: A randomized controlled study. Complement Ther Clin Pract. 2020 May;39:101166. doi: 10.1016/j.ctcp.2020.101166. Epub 2020 Apr 1. PMID 32379637
- [Result] Mendes LP, Moraes KS, Hoffman M, Vieira DS, Ribeiro-Samora GA, Lage SM, Britto RR, Parreira VF. Effects of Diaphragmatic Breathing With and Without Pursed-Lips Breathing in Subjects With COPD. Respir Care. 2019 Feb;64(2):136-144. doi: 10.4187/respcare.06319. Epub 2018 Aug 28. PMID 30154127
- [Result] Ubolnuar N, Tantisuwat A, Thaveeratitham P, Lertmaharit S, Kruapanich C, Mathiyakom W. Effects of Breathing Exercises in Patients With Chronic Obstructive Pulmonary Disease: Systematic Review and Meta-Analysis. Ann Rehabil Med. 2019 Aug;43(4):509-523. doi: 10.5535/arm.2019.43.4.509. Epub 2019 Aug 31. PMID 31499605